CLINICAL TRIAL: NCT00055237
Title: Phase II Study of Intravenous Recombinant Humanized Anti-Vascular Endothelial Cell Growth Factor Antibody (Bevacizumab) in Classical (HIV-Negative) and in AIDS-Associated Kaposi's Sarcoma
Brief Title: Bevacizumab to Treat Kaposi's Sarcoma in HIV-Positive and HIV-Negative Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Robert Yarchoan, Principal Investigator, National Institutes of Health Clinical Center (CC)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 030110; 03-C-0110; NCT00058136 (obsolete NCT alias)
Record Dates: First submitted 2003-02-21; First posted 2003-02-21 (Estimated); Results first posted 2012-07-26 (Estimated); Last update posted 2017-09-06 (Actual); Status verified 2017-08

CONDITIONS: Kaposi's Sarcoma; HIV Infections; HIV Seronegativity
Keywords: Angiogenesis; Cancer; HHV-8; KSHV; Skin; Kaposi Sarcoma; KS
MeSH Terms: conditions — Sarcoma, Kaposi; HIV Infections; Neoplasms | interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1: Pts with HIV-associated Kaposi's Sarcoma (Experimental): 15 mg/kg bevacizumab intravenously on days 1 and 8 then every 3 weeks.
  Interventions: Biological: Bevacizumab
- Cohort 2: Pts with classic Kaposi's Sarcoma (HIV-uninfected) (Experimental): 15 mg/kg bevacizumab intravenously on days 1 and 8 then every 3 weeks.
  Interventions: Biological: Bevacizumab

INTERVENTIONS:
Biological: Bevacizumab — 15 mg/kg day intravenously on day 1, day 8, then every 3 weeks.
  Other Names: Avastin

SUMMARY:
This study will examine the safety and effectiveness of the experimental drug bevacizumab for treating both non-acquired immune deficiency syndrome (AIDS) and AIDS-associated Kaposi's sarcoma (KS). KS tumors depend on the formation of new blood vessels for their growth. Bevacizumab is an antibody to a protein called vascular endothelial growth factor (VEGF) that is produced by the body and is involved in blood vessel growth. Bevacizumab may block the action of VEGF, and thus help shrink KS lesions.

Patients 18 years of age and older with Kaposi's sarcoma that is restricted to the skin and is not life threatening may be eligible for this study. Candidates will be screened with a medical history and physical examination, blood and urine tests, electrocardiogram (EKG), chest x-ray, and, if needed, imaging studies to evaluate internal tumors.

Participants will receive bevacizumab intravenously (by vein) once a week for 2 weeks and then every 3 weeks at the National Institutes of Health (NIH) Clinical Center. The first infusion takes about 90 minutes, the second takes about 60 minutes, and subsequent infusions take about 30 minutes. Infusions may take longer, however, if the drug is better tolerated at a slower infusion rate. Patients will be evaluated with the following tests and procedures:

* Physical examination, assessment of drug side effects, measurement of KS lesions, and photographs of lesions once a week for the first 6 weeks of therapy, and then every 3 weeks.
* cluster of differentiation 4 (CD4) cell counts and human immunodeficiency virus (HIV) viral load in HIV-positive patients every 12 weeks.
* Biopsies of lesions: upon entering the study, at week 12, and at the time of a response of the tumor to therapy or at the end of treatment, if treatment ends at week 18 or later.
* Additional biopsies, if requested. (Additional biopsies are not required.)
* Other procedures, such as computed tomography (CT) or magnetic resonance imaging (MRI) scans, if medically indicated.

Patients may continue bevacizumab therapy indefinitely if they are benefiting from it, as long as they have no substantial toxicity or other conditions that would cause them to stop receiving it and the protocol remains open.

DETAILED DESCRIPTION:
BACKGROUND:

This is a phase II study to determine the activity of bevacizumab, a putative antiangiogenic agent, in Kaposi's sarcoma (KS). Bevacizumab is a humanized recombinant antibody to vascular endothelial cell growth factor (VEGF), an important cytokine in the pathogenesis of KS.

OBJECTIVES:

To assess the antitumor effect of bevacizumab 15 mg/kg administered intravenously once every three weeks in patients with human immunodeficiency virus (HIV)-associated Kaposi's sarcoma (KS). Other objectives include assessment of the antitumor effect of bevacizumab 15 mg/kg administered intravenously once every three weeks in patients with classical KS; assessment of the toxicity profile of bevacizumab in HIV-infected and HIV-negative patients with KS; exploration in a preliminary fashion effect of bevacizumab on KS progression free survival; and study of a number of biochemical parameters, including stromal cell-derived factor-1 (SDF-1) expression in KS lesions; human herpes virus-8 (HHV-8) viral load in peripheral blood mononuclear cells; serum vascular endothelial growth factor (VEGF) levels over the course of treatment; and changes in viral interleukin 6 (IL-6) levels over the course of treatment.

ELIGIBILITY:

Key eligibility parameters include HIV-associated or classical Kaposi's sarcoma, age greater than or equal to 18 years, and life expectancy greater than 6 months. Patients with HIV infection must have either KS progression on a regimen of highly active antiretroviral therapy (HAART) for at least one month, or no KS regression while on an optimized regimen of HAART for 4 months or longer.

DESIGN:

Patients will be sequentially enrolled, administered a loading dose of 15 mg/kg bevacizumab intravenously on day 1, and then administered 15 mg/kg bevacizumab intravenously every 3 weeks beginning one week after the loading dose. The drug will be temporarily discontinued for toxicity, intercurrent major surgical procedures, or other factors that would pose a safety concern. Patients will undergo a biopsy of a KS lesion at entry, on cycle 4, day 21, and at the time of a formal response or when the patient stops treatment. Patients will undergo a number of other tests as well, including blood tests and non-invasive imaging studies of KS lesions.

ELIGIBILITY:
* INCLUSION CRITERIA:

Age greater than or equal to 18 years.

Kaposi's sarcoma pathologically confirmed by Center for Cancer Research (CCR) pathology.

Eastern Cooperative Oncology Group (ECOG) performance status less than or equal to 2.

Life expectancy greater than 6 months.

The following hematologic parameters:

* Hemoglobin greater than 9 g/dl;
* White blood cell (WBC) greater than 1000/mm^3;
* Absolute neutrophil count (ANC) greater than 750/mm^3;
* Platelets greater than 75,000/mm^3;
* Prothrombin time (PT) and partial thromboplastin time (PTT) less than or equal to 120% of control, unless patient has the presence of a lupus anticoagulant.

The following hepatic parameters:

Bilirubin less than or equal to 1.5 times the upper limit of normal (ULN) unless the patient is receiving protease inhibitor therapy known to be associated with increased bilirubin:

in this case total bilirubin less than or equal to 7.5 mg/dl and the direct fraction less than or equal to 0.7 mg/dl.

-Examples of protease inhibitors known to increase bilirubin levels include indinavir, ritonavir, nelfinavir, and atazanavir.

Aspartate aminotransferase (AST)/glutamic oxaloacetic transaminase (GOT) less than or equal to 2.5 times the upper limit of normal.

Either Serum creatinine less than or equal to 1.5 mg/dL or measured creatinine clearance greater than or equal to 60 mL/min.

Either Urine protein less than 1+ or measured 24 hour urine protein less than 500 milligram.

Blood pressure: systolic blood pressure (SBP) less than 160 mm/Hg; diastolic blood pressure (DBP) less than 95 mm/Hg.

At least 5 assessable cutaneous lesions previously untreated by local therapy.

Patients with human immunodeficiency virus (HIV) infection must be willing to comply with a regimen of highly active antiretroviral therapy and be on a regimen of highly active antiretroviral therapy (HAART) selected for best potential efficacy for at least 1 month with evidence of Kaposi sarcoma (KS) progression on the HAART regimen or be on a optimized regimen of HAART for 4 months or longer with no evidence of KS regression.

Patients must be willing to use effective birth control.

EXCLUSION CRITERIA:

Symptomatic, extensive pulmonary involvement.

Symptomatic visceral KS excluding the oral cavity.

Inability to provide informed consent.

Chemotherapy within 3 weeks.

Prior therapy with SU5416.

Supraphysiologic doses of corticosteroids within 3 weeks.

Major surgical procedure (including periodontal) within 4 weeks.

Surgical or other non-healing wounds unrelated to KS.

Pregnancy.

Breast feeding.

Past or present history of malignant tumors other than KS unless: a) in a complete remission for greater than or equal to 1 year from the time a response was first documented; b) completely resected basal cell carcinoma; or c) in situ squamous cell carcinoma of the cervix or anus.

Evidence of a severe or life-threatening infection within 2 weeks of entry onto the study.

A condition that would require the patient to receive intravenous antibiotics on a day of bevacizumab infusion.

Need for chronic daily aspirin greater than or equal to 325 mg/daily or nonsteroidal medication interfering with platelet function.

Therapeutic anticoagulation with international normalized ratio (INR) greater than 1.5, unless the patient is on full dose warfarin. If a patient is on full-dose anticoagulants, the following criteria should be met for enrollment:

The subject must have an in-range INR (usually between 2 and 3) on a stable dose of warfarin or on stable dose of low molecular weight (LMW) heparin;

The subject must not have active bleeding or pathological conditions that carry high risk of bleeding (e.g. tumor involving major vessels).

History of deep venous or arterial thrombosis.

History of gastrointestinal bleeding.

Clinically significant cardiovascular disease such as uncontrolled hypertension (with systolic BP greater than 160 mm/Hg or diastolic blood pressure greater than 95 mm/Hg), unstable angina, New York Heart Association grade II or greater congestive heart failure, cardiac arrhythmia requiring medication, clinically significant peripheral artery disease, grade II or greater peripheral vascular disease, myocardial infarction.

Substantial central nervous system (CNS) disease including history of CNS bleeding, mass lesions in the brain, uncontrolled seizure disorder, recent history of cerebrovascular accident (CVA) (e.g. within the past 6 months), history of transient ischemic attack (TIA) within the past 6 months..

Coagulopathy.

Patients with unstable bone fractures that are not stress/weight bearing able.

Patients with any other abnormality that would be scored as a grade 3 toxicity, except lymphopenia, direct manifestations of KS, direct manifestation of HIV, direct manifestation of HIV therapy, hyperbilirubinemia associated with protease inhibitors, asymptomatic hyperuricemia.

Previous intravenous immunoglobulin (IVIG) or monoclonal antibody therapy within 30 days prior to enrollment.

Known hypersensitivity to bevacizumab.

Known hypersensitivity to Chinese hamster ovary cell products.

Known hypersensitivity to other recombinant human or humanized antibodies.

Previous bevacizumab.

Any condition that, in the opinion of the Principal Investigator or Study Chairperson, would preclude the inclusion of a patient onto this research study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2003-02-26 (Actual); Primary Completion 2010-03-15 (Actual); Study Completion 2010-03-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Yarchoan, M.D., Principal Investigator — National Cancer Institute, National Institutes of Health
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Uldrick TS, Wyvill KM, Kumar P, O'Mahony D, Bernstein W, Aleman K, Polizzotto MN, Steinberg SM, Pittaluga S, Marshall V, Whitby D, Little RF, Yarchoan R. Phase II study of bevacizumab in patients with HIV-associated Kaposi's sarcoma receiving antiretroviral therapy. J Clin Oncol. 2012 May 1;30(13):1476-83. doi: 10.1200/JCO.2011.39.6853. Epub 2012 Mar 19. PMID 22430271
- [Result] Uldrick T, Wyvill K, Kumar P, Bernstein W, O'Mahony D, Polizzotto M, Aleman K, Steinberg S, Pittaluga S, Little R, and Yarchoan R. A Phase II Study Targeting Vascular Endothelial Growth Factor with the Humanized Monoclonal Antibody Bevacizumab in the Treatment of Patients with HIV-Associated Kaposi Sarcoma. 17th Conference on Retroviruses and Opportunistic Infections. Oral Presentation. February 17, 2010.

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1: Cohort 1: Pts With HIV-associated Kaposi's Sarcoma; Cohort 2: Pts With Classic Kaposi's Sarcoma (HIV-uninfected): 15 mg/kg bevacizumab intravenously on days 1 and 8 then every 3 weeks
Period: Overall Study
Arm/Group | Cohort 1: Cohort 1: Pts With HIV-associated Kaposi's Sarcoma | Cohort 2: Pts With Classic Kaposi's Sarcoma (HIV-uninfected)
Started | 17 | 2
Completed | 17 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: Cohort 1: Pts With HIV-associated Kaposi's Sarcoma | Cohort 2: Pts With Classic Kaposi's Sarcoma (HIV-uninfected) | Total
Number analyzed (Participants) | 17 | 2 | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 2 | 17
  >=65 years | 2 | 0 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 42 (9.3) | 58 (12.7) | 50 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 16 | 2 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic | 3 | 0 | 3
  Not Hispanic or Latino | 14 | 2 | 16
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 17 | 2 | 19

OUTCOME MEASURES:

1. Primary Outcome: Response Rate
Description: Percentage of participants with a complete response (CR) + partial response (PR)per the Modified AIDS Clinical Trial Group Criteria (ACTG) for HIV-KS. PR is a 50% decrease in the number and/or size of previously existing lesions for 4 weeks; or complete flattening of at least 50% of all previously raised lesions lasting for at least 4 weeks; or a 50% decrease in the sum of the products of the largest perpendicular diameters of the marker lesions lasting for at least 4 weeks; CR is the absence of any detectable residual disease, including tumor associated edema, persisting for at least 4 weeks.
Time Frame: 36 months
Population: Cohort 2 is not reported here because response rate in HIV negative patients was a secondary outcome.
Measure: Mean (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 1: Cohort 1: Pts With HIV-associated Kaposi's Sarcoma
Number analyzed (Participants) | 16
Percentage of participants | 31 [11 to 58.7]
Statistical Analysis 1: Comparison: Cohort 1: Cohort 1: Pts With HIV-associated Kaposi's Sarcoma; Test type: Superiority or Other; sample estimate with 95% CI; proportion estimate,binomial exact 95%CI = 31, 95% CI 2-sided [11 to 58.7], Standard Deviation 11.6 — As stated in the Outcome statistical Analysis 1. Section, the confidence interval was calculated using binomial exact statistics. The standard deviation is based on that calculation

2. Secondary Outcome: Number of Participants With Adverse Events
Description: Here are the number of participants with adverse events. For the detailed list of adverse events, see the adverse event module.
Time Frame: 70 months
Population: All adverse events regardless of attribution, over 202 cycles in 19 patients. Per protocol analysis of adverse events.
  Cohort 1 and 2 are reported together.
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 1 & 2: Pts With HIV-associated and Classic KS: 15 mg/kg bevacizumab intravenously on days 1 and 8 then every 3 weeks
Arm/Group | Cohort 1 & 2: Pts With HIV-associated and Classic KS
Number analyzed (Participants) | 19
Participants | 19

ADVERSE EVENTS:
Time Frame: 70 months
Arm/Group | Cohort 1 & 2: Pts With HIV-associated and Classic KS
All-Cause Mortality (participants affected / at risk) | 0/19
Serious Adverse Events (participants affected / at risk) | 4/19
Other Adverse Events (participants affected / at risk) | 19/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 & 2: Pts With HIV-associated and Classic KS (N=19)
Acidosis (metabolic or respiratory) (Metabolism and nutrition disorders) | 1 (1)
Adult respiratory distress syndrome (ARDS) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bicarbonate (Investigations) | 1 (1)
CPK (creatine phosphokinase) (Investigations) | 1 (1)
Creatinine (Investigations) | 1 (1)
Hemoglobin (Investigations) | 1 (3)
Hypotension (Vascular disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Infection (Infections and infestations) | 1 (1) — (documented clinically or microbiologically) with grade 3 or 4 neutropenia (ANC <1.0 x 10e
Infection/Febrile Neutropenia-Other (Specify, from leg cellulitis) (Infections and infestations) | 3 (3)
Partial thromboplastin time (PTT) (Investigations) | 1 (1)
Platelets (Investigations) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1)
Syndromes-Other (Specify, toxic shock syndrome) (General disorders) | 1 (1)
Transfusion: Platelets (Blood and lymphatic system disorders) | 1 (1)
Vomit (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 & 2: Pts With HIV-associated and Classic KS (N=19)
Abdominal pain or cramping (Gastrointestinal disorders) | 1 (1)
Alkaline phosphatase (Investigations) | 2 (8)
Allergic rhinitis (including sneezing, nasal stuffiness, postnasal drip) (Immune system disorders) | 8 (10)
Amylase (Investigations) | 9 (20)
Anorexia (Gastrointestinal disorders) | 2 (2)
Bilirubin (Investigations) | 11 (26)
CPK (creatine phosphokinase) (Investigations) | 8 (27)
Constipation (Gastrointestinal disorders) | 5 (6)
Cough (Respiratory, thoracic and mediastinal disorders) | 9 (15)
Creatinine (Investigations) | 3 (6)
Dermatology/Skin-Other (Specify, foot callous; burning sensation in abdominal area) (Skin and subcutaneous tissue disorders) | 2 (2)
Diarrhea patients without colostomy (Gastrointestinal disorders) | 9 (17)
Dizziness/lightheadedness (Nervous system disorders) | 2 (2)
Dry eye (Eye disorders) | 1 (1)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dysuria (painful urination) (Renal and urinary disorders) | 1 (1)
Edema (General disorders) | 3 (5)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 8 (12)
Fatigue (lethargy, malaise, asthenia) (General disorders) | 5 (9)
Fever (General disorders) | 9 (13) — (in the absence of neutropenia, where neutropenia is defined as AGC<1.0 x 10e9/L)
Gastrointestinal-Other (Specify, bloating fullness; slight indigestion) (Gastrointestinal disorders) | 2 (2)
Headache (Nervous system disorders) | 11 (30)
Hematuria (in the absence of vaginal bleeding) (Renal and urinary disorders) | 8 (10)
Hemoglobin (Investigations) | 10 (31)
Hemoglobinuria (Renal and urinary disorders) | 10 (23)
Hemolysis (e.g., immune hemolytic anemia, drug related hemolysis, other) (Blood and lymphatic system disorders) | 1 (2)
Hemorrhage-Other (Specify, gums; gums bleeding) (Blood and lymphatic system disorders) | 1 (2)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1)
Hypercholesterolemia (Metabolism and nutrition disorders) | 3 (4)
Hyperglycemia (Metabolism and nutrition disorders) | 8 (37)
Hyperkalemia (Metabolism and nutrition disorders) | 2 (2)
Hypermagnesemia (Metabolism and nutrition disorders) | 4 (8)
Hypertension (Vascular disorders) | 10 (18)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 3 (7)
Hyperuricemia (Metabolism and nutrition disorders) | 3 (10)
Hypoalbuminemia (Metabolism and nutrition disorders) | 13 (48)
Hypocalcemia (Metabolism and nutrition disorders) | 7 (25)
Hypoglycemia (Metabolism and nutrition disorders) | 5 (8)
Hypokalemia (Metabolism and nutrition disorders) | 2 (9)
Hypomagnesemia (Metabolism and nutrition disorders) | 8 (17)
Hyponatremia (Metabolism and nutrition disorders) | 12 (46)
Hypophosphatemia (Metabolism and nutrition disorders) | 8 (21)
Hypothyroidism (Endocrine disorders) | 1 (1)
Infection without neutropenia (Infections and infestations) | 3 (5)
Infection/Febrile Neutropenia-Other (Specify) (Infections and infestations) | 2 (4) — fungal infections, feet tinea pedis; URI; swelling behind R knee; tinea L axilla
Insomnia (Psychiatric disorders) | 3 (4)
Leukocytes (total WBC) (Investigations) | 8 (33)
Lipase (Investigations) | 3 (7)
Lymphopenia (Investigations) | 4 (11)
Mouth dryness (Gastrointestinal disorders) | 1 (1)
Musculoskeletal-Other (Specify, joint stiffness) (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (muscle pain) (Musculoskeletal and connective tissue disorders) | 5 (8)
Nausea (Gastrointestinal disorders) | 6 (7)
Neuropathy-sensory (Nervous system disorders) | 4 (6)
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 1 (1) — for leukemia studies or bone marrow infiltrative/myelophthisic process, if specified in the protocol.
Pain-Other (back pain;leg pain; heel pain; throat pain; from leg cellulitis; in R posterior knee) (General disorders) | 10 (27) — continued plantar fascilitis;jaw pain;knee pain;local pain foot/leg;pressure R mid back;sore throat;tooth pain;burn L thumb;chest pain;cramps in feet;soreness L index finger;knee-tumor pain;leg pain;side mandibular LN tender; infection,abcess tooth
Palpitations (Cardiac disorders) | 1 (1)
Partial thromboplastin time (PTT) (Investigations) | 10 (16)
Pigmentation changes (e.g., vitiligo) (Skin and subcutaneous tissue disorders) | 1 (1)
Platelets (Blood and lymphatic system disorders) | 11 (25)
Proteinuria (Renal and urinary disorders) | 14 (56)
Prothrombin time (PT) (Investigations) | 6 (10)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (3)
Pulmonary-Other (Specify, sneezing) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 4 (7)
Rectal bleeding/hematochezia (Gastrointestinal disorders) | 1 (1)
Rigors, chills (General disorders) | 2 (2)
SGOT (AST) (serum glutamic oxaloacetic transaminase) (Investigations) | 13 (45)
SGPT (ALT) (serum glutamic pyruvic transaminase) (Investigations) | 8 (22)
Sweating (diaphoresis) (Skin and subcutaneous tissue disorders) | 5 (5)
Taste disturbance (dysgeusia) (Nervous system disorders) | 2 (2)
Tumor pain (onset or exacerbation of tumor pain due to treatment) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Vision-blurred vision (Eye disorders) | 1 (1)
Vision-flashing lights/floaters (Eye disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 6 (7)
Weight loss (Investigations) | 2 (2)
Arthralgia (joint pain) (Musculoskeletal and connective tissue disorders) | 4 (7)
Cardiac left ventricular function (Cardiac disorders) | 1 (1)
Cardiac troponin I (cTnI) (Cardiac disorders) | 1 (1)
CD4 count (Investigations) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Gynecomastia (Reproductive system and breast disorders) | 1 (1)
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 13 (54) — Neutrophils/granulocytes (ANC/AGC) for leukemia studies or bone marrow infiltrative/myelophthisic process, if specified in the protocol.
Phlebitis (superficial) (Vascular disorders) | 1 (1)
Thrombosis/embolism (Vascular disorders) | 1 (1)
Vaginal bleeding (Reproductive system and breast disorders) | 1 (1)
Auditory/Hearing-Other (Specify, hearing loss) (Ear and labyrinth disorders) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1)
Nail changes (Skin and subcutaneous tissue disorders) | 1 (1)
Neuropathy - cranial (Nervous system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No